CLINICAL TRIAL: NCT01885715
Title: Appropriate Dose of Neostigmine for Reversal of Rocuronium and Cisatracurium
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B-1208/168-009; Eunsu Choi (Registry Identifier: Eunsu Choi)
Record Dates: First submitted 2013-06-14; First posted 2013-06-25 (Estimated); Last update posted 2014-06-13 (Estimated); Status verified 2014-06

CONDITIONS: Observation of Neuromuscular Block

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (8):
- Rocuronium-placebo (Placebo Comparator): At anesthetic induction, rocuronium 0.6 mg/kg will be injected for muscle relaxation.
  During surgical procedure, we will monitor train of four (TOF) using nerve stimulator. When TOF ratio recover to 0.5, normal saline 5 ml will be injected. And we will measure time to take from TOF ratio 0.5 to 1.0
  Interventions: Drug: Injection of neostigmine
- Rocuronium-neostigmine 10 ㎍ (Active Comparator): At anesthetic induction, rocuronium 0.6 mg/kg will be injected for muscle relaxation.
  During surgical procedure, we will monitor train of four(TOF)using nerve stimulator. When TOF ratio recover to 0.5, neostigmine 10 ㎍/kg will be injected. And we will measure time to take from TOF ratio 0.5 to 1.0.
  Interventions: Drug: Injection of neostigmine
- Rocuronium-neostigmine 20 ㎍ (Active Comparator): At anesthetic induction, rocuronium 0.6 mg/kg will be injected for muscle relaxation.
  During surgical procedure, we will monitor train of four(TOF)using nerve stimulator. When TOF ratio recover to 0.5, neostigmine 20 ㎍/kg will be injected. And we will measure time to take from TOF ratio 0.5 to 1.0
  Interventions: Drug: Injection of neostigmine
- Rocuronium-neostigmine 40 ㎍ (Active Comparator): At anesthetic induction, rocuronium 0.6 mg/kg will be injected for muscle relaxation.
  During surgical procedure, we will monitor train of four(TOF)using nerve stimulator. When TOF ratio recover to 0.5, neostigmine 40 ㎍/kg will be injected. And we will measure time to take from TOF ratio 0.5 to 1.0
  Interventions: Drug: Injection of neostigmine
- Cisatracurium-placebo (Placebo Comparator): At anesthetic induction, cisatracurium 0.15 mg/kg will be injected for muscle relaxation.
  During surgical procedure, we will monitor train of four(TOF)using nerve stimulator. When TOF ratio recover to 0.5, normal saline 5 ml will be injected. And we will measure time to take from TOF ratio 0.5 to 1.0
  Interventions: Drug: Injection of neostigmine
- Cisatracurium-neostigmine 10 ㎍ (Active Comparator): At anesthetic induction, cisatracurium 0.15 mg/kg will be injected for muscle relaxation.
  During surgical procedure, we will monitor train of four(TOF)using nerve stimulator. When TOF ratio recover to 0.5, neostigmine 10 ㎍/kg will be injected. And we will measure time to take from TOF ratio 0.5 to 1.0
  Interventions: Drug: Injection of neostigmine
- Cisatracurium-neostigmine 20 ㎍ (Active Comparator): At anesthetic induction, cisatracurium 0.15 mg/kg will be injected for muscle relaxation.
  During surgical procedure, we will monitor train of four(TOF)using nerve stimulator. When TOF ratio recover to 0.5, neostigmine 20 ㎍/kg will be injected. And we will measure time to take from TOF ratio 0.5 to 1.0
  Interventions: Drug: Injection of neostigmine
- Cisatracurium-neostigmine 40 ㎍ (Active Comparator): At anesthetic induction, cisatracurium 0.15 mg/kg will be injected for muscle relaxation.
  During surgical procedure, we will monitor train of four(TOF)using nerve stimulator. When TOF ratio recover to 0.5, neostigmine 40 ㎍/kg will be injected. And we will measure time to take from TOF ratio 0.5 to 1.0
  Interventions: Drug: Injection of neostigmine

INTERVENTIONS:
Drug: Injection of neostigmine — At induction, we will inject rocuronium 0.6 mg/kg for rocuronium arms and cisatracurium 0.15 mg/kg for cisatracurium arms.
  During surgical procedure, we will monitor train of four(TOF)using nerve stimulator. When TOF ratio recover to 0.5, normal saline 5 ml will be injected in placebo arms. And neostigmine 10, 20, or 40 ㎍/kg will injected in each arms.

SUMMARY:
This study aims to find appropriate dose of neostigmine which is possible to reverse rocuronium or cisatracurium till train of four (TOF) 0.9 within 10 minutes.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist Physical status classification 1 or 2 elective surgery under general anesthesia

Exclusion Criteria:

* BMI >25 or < 20 kg/m2
* Patients taking intercurrent medication
* Glutamic Oxalacetate Transaminase or Glutamic Pyruvate Transaminase > 40 IU/L, Cr > 1.4 mg/dl

Ages: 19 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2013-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
time to reverse from light muscle relaxation | time from TOF 0.5 to TOF 1.0 after injection of different doses of neostigmine
  Primary outcome of this study is how long it takes time to reverse from TOF ratio 0.5 to 1.0 after injection of different doses of neostigmine at the TOF 0.5

SECONDARY OUTCOMES:
time to reverse from TOF ratio 0.5 to 0.9 | time from TOF 0.5 to TOF 0.9 after injection of different doses of neostigmine
  Secondary outcome of this study is how long it takes time to reverse from TOF ratio 0.5 to 0.9 after injection of different doses of neostigmine at the TOF 0.5

CONTACTS AND LOCATIONS:
Overall Officials: Ah Young Oh, Principal Investigator — Professor
Locations (1):
- Eunsu Choi, Seongnam-si, Gyeonggi-do, South Korea